CLINICAL TRIAL: NCT03954912
Title: Comparative Outcomes Between Image-based (MAKO) Versus Imageless NAVIO Robot-assisted Unicondylar Knee Arthroplasty
Brief Title: Comparative Outcomes Between Image-based Versus Imageless Robot-assisted Unicondylar Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Bhumibol Adulyadej Hospital (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/62
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee
Keywords: MAKO; NAVIO; robotic surgery; UKA; surgical time; KSS; KFS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MAKO robotic assisted UKA (Active Comparator): image base (MAKO) robotic assisted UKA
  Interventions: Procedure: MAKO assisted unicondylar knee arthroplasty
- NAVIO robotic assisted UKA (Active Comparator): imageless (NAVIO) robotic assisted UKA
  Interventions: Procedure: NAVIO assisted unicondylar knee arthroplasty

INTERVENTIONS:
Procedure: MAKO assisted unicondylar knee arthroplasty — MAKO assisted
  Arms: MAKO robotic assisted UKA
Procedure: NAVIO assisted unicondylar knee arthroplasty — NAVIO assisted
  Arms: NAVIO robotic assisted UKA

SUMMARY:
This prospective cohort study was conducted with the aim of comparing relevant clinical outcomes which included intra (surgical time and blood loss), post-operative outcomes (range of motion, function, complications and revisions) and return to activity between imageless and image-based surgical system in medial unicondylar knee arthroplasty

DETAILED DESCRIPTION:
this prospective cohort study was conducted between 1st June 2015 and 1st July 2018 at Bhumibol Adulyadej Hospital, Bangkok, Thailand. A total of 33 medial compartment OA knee patients were randomly allocated to MAKO or NAVIO robotic assisted UKA. The outcomes assessed were intra-operative outcomes (operative time, blood loss) and postoperative outcomes (function, complications and revision) at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients were those deemed suitable for unicondylar knee arthroplasty surgery
* patients who could give informed consent
* patients who willing to attend the prescribed follow-up.

Exclusion Criteria:

* Patients who have medial osteoarthritis knee with following condition:

  1. Ligament insufficiency (anterior cruciate ligament rupture, collateral ligament insufficiency).
  2. Inflammatory arthritis
  3. A deformity requiring augmentation
  4. Neurological movement disorders
  5. pathology of the feet, ankles, hips, or opposite knee causing significant pain or gait alterations
* Patients who ultimately required a total knee arthroplasty (valgus greater than 14 degree, multiple compartment osteoarthritis were contraindications to unicondylar knee arthroplasty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
operative time | 1 day
  operative time in minutes the higher value of blood loss is worse outcome
calculated total blood loss | 1 day
  total blood loss which was calculated using a formula based on patient blood volume and a decrease in hemoglobin

SECONDARY OUTCOMES:
post operative complications | 12 months
  post operative complications included infection, wound complication, stiffness and revision. the higher number of post operative outcome is the worse outcomes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leelasestaporn C, Tarnpichprasert T, Arirachakaran A, Kongtharvonskul J. Comparison of 1-year outcomes between MAKO versus NAVIO robot-assisted medial UKA: nonrandomized, prospective, comparative study. Knee Surg Relat Res. 2020 Mar 12;32(1):13. doi: 10.1186/s43019-020-00030-x. PMID 32660619